CLINICAL TRIAL: NCT05816772
Title: Comparison of Post-Operative Pain After Use of Calcium Hydroxide and Bio Ceramic Sealer for Root Canal Treatment: A Randomized Clinical Trial.
Brief Title: Comparison of Post-Operative Pain After Use of Calcium Hydroxide and Bio Ceramic Sealer for Root Canal Treatment.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, syed hasan shaharyar, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HShaharyar
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endosequence Bio ceramic based Sealer (Experimental): Sealer was introduced into the canal by coating the master gutta-percha point (Endosequence, Brasseler USA, Gutta Percha ) with sealer, followed by cold lateral compaction using a finger spreader # 30 and # 35 (Saybron Endo) with decreasing working length by 1-2 mm. A heated plugger was used to sear off GuttaPercha coronal to canal orifice.Recordings of postoperative pain was obtained at 24 hours, 48 hours, 72 hours and 7 days after obturation with aid of the Visual Analogue Scale.
  Interventions: Drug: Endosequence Bio ceramic Sealer
- Sealapex calcium hydroxide based sealer (Active Comparator): Sealer was introduced into the canal by coating the master gutta-percha point (Dentsply Sirona, GuttaPercha Conform fit) with sealer, followed by cold lateral compaction using a finger spreader # 30 and # 35 (Saybron Endo) with decreasing working length by 1-2 mm. A heated plugger was used to sear off GuttaPercha coronal to canal orifice.Recordings of postoperative pain was obtained at 24 hours, 48 hours, 72 hours and 7 days after obturation with aid of the Visual Analogue Scale.
  Interventions: Drug: Sealapex Calcium hydroxide Based Sealer

INTERVENTIONS:
Drug: Endosequence Bio ceramic Sealer — Brasseler,USA, a nano-particulate injectable premixed bioceramic sealer that contains Calcium Silicates, Calcium Phosphate, Calcium Hydroxide and Zirconium Oxide
  Arms: Endosequence Bio ceramic based Sealer
Drug: Sealapex Calcium hydroxide Based Sealer — KERR Dental, an original eugenol-free root canal sealant based on calcium hydroxide.
  Arms: Sealapex calcium hydroxide based sealer

SUMMARY:
Background:

Root canal therapy is a well documented and established method to eliminate inflamed pulp and reduce pain, but the procedure itself is associated with postoperative discomfort, ranging from 1.2%-82.9% in different studies. There are several treatment-related factors that are found to be linked to postoperative pain, including gauging canal length with apex locator, the choice of instrumentation, number of visits and the root canal sealer being used. When used in the root canal obturation, an endodontic sealer may affect periodontal tissue through apical foramina, lateral canals, or leaching and can hinder the healing process. Thus, the local inflammation caused by root canal obturation may result in post-operative pain. The extent of inflammatory response depends on multiple factors, which also include the content of the sealer.

The reason of using calcium hydroxide sealers is driven by their potential for tissue healing and antibacterial properties. Antimicrobial effects of Calcium Hydroxide is attributed to the presences and numbers of hydroxyl groups which cause pH to increase as high as 12.5.

The elevated pH levels also encourage repair and bone ossification, thus helping in healing. Hard tissue formation which is associated with calcium hydroxide's alkaline nature occurs due to inhibition of lactic acid secreted by osteoclast, activation of Alkaline phosphatase and calcium-dependent ATP.

Bioceramic sealers are considered to provide better results for root canals treatments by promoting osteoblastic differentiation and by releasing bioactive substances. Cytotoxicity of bioceramics is lower in comparision of resin-based sealers. Less cytotoxicity also lowers the potential of irritation and inflammation of periodontal tissues, thus leading to reduced levels of associated post-operative pain. Very limited data is available on the comparison between calcium hydroxide and bioceramic sealer.

Objectives:

1. To compare pre and postoperative pain within each group(calcium hydroxide sealer and Bioceramic sealer).
2. Compare postoperative pain between calcium hydroxide sealer and Bioceramic sealer groups.
3. To observe the effect of type of tooth and patient demographics on postoperative pain in each group.

Methods:

After taking consent, A total of 80 patients with symptomatic irreversible pulpitis will be randomly assigned to one of two groups in this 6-month In-Vitro Single-Blinded Randomized Clinical Study. Group A will receive calcium hydroxide as an endodontic sealer and B will receive bioceramic sealer respectively. Recordings of postoperative pain will be obtained at 24 hours, 48 hours, 72 hours and 7 days after obturation with aid of the Visual Analogue Scale by the Researcher.

SPSSv.24 will be used to analyze the data with the level of significance set at p < 0.05. For comparison of VAS scores, Paired Sample t-test//Wilcoxon-signed rank test will be used. Independent sample-test/Mann-Whitney U-test will be used to assess the differences in VAS pain scores between the groups. The chi-square test will be used to determine the frequency of tooth types among the tested materials and the distribution of patients among VAS scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need root canal treatment of minimum one tooth.
* Patients between 18 years to 60 years of age.
* Single rooted tooth with a single (type I canal configuration according to vertucci) canal including mandibular and maxillary incisors, canine and premolars except maxillary first premolar.
* Tooth is diagnosed with symptomatic Irreversible Pulpitis.
* The periapical index score is from 2 to 3 according to Orstavik et al.

Exclusion Criteria:

* • Medically compromised patients.

  * Patient rejecting to participate in study.
  * Inability to achieve the full length of canal.
  * Teeth with periodontal disease (probing depth >4mm).
  * Complication during treatment (separation of file, ledge formation, etc.).
  * Pulpal necrosis, chronic apical periodontitis, acute and chronic periodontal abcess.
  * Any swelling or draining sinus.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Comparison of Post-Operative Pain After Use of Calcium Hydroxide and Bio Ceramic Sealer for Root Canal Treatment. | Before application of experimental agents (Day 0)
  Comparison of postoperative pain assessed with the help of Visual Analog Scale(VAS). Recording was obtained at Day 0 before the application of experimental agents.
  Visual Analog Scale which will be scored as 0 (No Pain), 1-3 (Mild Pain), 4-6 (Moderate pain) and 7-10 ( Severe pain)
Comparison of Post-Operative Pain After Use of Calcium Hydroxide and Bio Ceramic Sealer for Root Canal Treatment. | 24 hour after application of experimental agents
  Comparison of postoperative pain assessed with the help of Visual Analog Scale(VAS). Recording was obtained at 24 hour after the application of experimental agents.
Comparison of Post-Operative Pain After Use of Calcium Hydroxide and Bio Ceramic Sealer for Root Canal Treatment. | 48 hour after application of experimental agents
  Comparison of postoperative pain assessed with the help of Visual Analog Scale(VAS). Recording was obtained at 48 hour after the application of experimental agents.
Comparison of Post-Operative Pain After Use of Calcium Hydroxide and Bio Ceramic Sealer for Root Canal Treatment. | 72 hour after application of experimental agents
  Comparison of postoperative pain assessed with the help of Visual Analog Scale(VAS). Recording was obtained at 72 hour after the application of experimental agents.
Comparison of Post-Operative Pain After Use of Calcium Hydroxide and Bio Ceramic Sealer for Root Canal Treatment. | 7 Days after application of experimental agents
  Comparison of postoperative pain assessed with the help of Visual Analog Scale(VAS). Recording was obtained at 7 Days after the application of experimental agents.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Hasan Shaharyar, BDS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow International Dental College (Defence campus), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No